CLINICAL TRIAL: NCT06159920
Title: Evaluation of the Diagnostic and Prognostic Role of PET (PET/CT and PET/MRI) in Neuroendocrin Tumors.
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PET-NET-Retrospective
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: diagnostic accuracy — The aim of this retrospective study is to evaluate the diagnostic and prognostic value of PET/MRI and PET/CT with the use of different radiopharmaceuticals (68Ga-DOTATOC -edotreotide, and 18F-FDG - fluorodeoxyglucose) for the study of patients suffering from neuroendocrine tumors. To this end, both traditional imaging parameters and the contribution of radiomic features will be investigated. The latter are quantitative features extracted from biomedical images, and are believed to be able to provide information, otherwise impossible to investigate, useful for the characterization of various pathologies.

SUMMARY:
Neuroendocrine tumors (NETs) constitute approximately 0.5% of malignancies. To date, diagnosis at an increasingly early stage of the disease is possible thanks to recent technological advances in biomedical imaging. In particular, the traditional work-up for these pathologies includes endoscopy, magnetic resonance imaging (MRI) and computed tomography (CT). Furthermore, the integrated positron emission tomography methods (PET/CT and PET/MRI) are innovative molecular imaging techniques and represent a continually expanding field of research in the oncology setting. In particular, PET is taking on an increasingly relevant role for the study of neuroendocrine tumors, also thanks to the introduction of increasingly accurate radiopharmaceuticals (targeted towards somatostatin receptors), thus opening the way to new possibilities for the diagnosis andcharacterization of these tumors, is in the staging and restaging phase .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients affected by neuroendocrine tumors; Patients who have performed at least one PET study with 18F-FDG and/or 68Ga- DOTATOC for the staging or diagnosis of their pathology.

Exclusion Criteria:

* Patients < 18 years old;
* Lack of availability of clinical data and PET imaging useful for analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, adult patients suffering from neuroendocrine tumors who have undergone PET examination (PET/CT or PET/MRI) with 18F-FDG or 68Ga-DOTATOC at the U.0 of Nuclear medicine at the RCCS San Raffaele will be considered for clinical reasons both in the staging and restaging phases.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2024-12-27 (Estimated)

PRIMARY OUTCOMES:
800 patients suffering from neuroendocrine tumors who have undergone PET examination (PET/CT or PET/MRI) with 18F-FDG or 68Ga-DOTATOC. | 2 years
  The integrated positron emission tomography methods (PET/CT and PET/MRI) are innovative molecular imaging techniques, for the diagnosis and characterization of these tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No